CLINICAL TRIAL: NCT00553748
Title: A Phase I, Open Label, Single Center Safety Study of [F-18]FLT
Brief Title: Phase I, Open Label, Single Center Safety Study of [F-18]FLT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Siemens Molecular Imaging (Industry)
Responsible Party: Charles Intenzo, MD, Thomas Jefferson University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: D0008186
Record Dates: First submitted 2007-11-02; First posted 2007-11-06 (Estimated); Last update posted 2008-07-03 (Estimated); Status verified 2008-07

CONDITIONS: Brain Cancer
MeSH Terms: conditions — Brain Neoplasms | interventions — alovudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- I (Experimental)
  Interventions: Drug: F-18 FLT

INTERVENTIONS:
Drug: F-18 FLT — One - 10 mci dose of F-18 FLT is administered IV over about 5 seconds prior to PET imaging. Each imaging dose contains no more than 6.1 micrograms of FLT.
  Other Names: 18-F FLT; [F-18]FLT

SUMMARY:
This is a ten subject, phase 1 study. The purpose of the Phase 1 study is to demonstrate drug safety in a target group of subjects with high grade brain cancer. This population represents a potential clinical population that may benefit from this PET imaging tracer. The study will also begin collection of baseline imaging data and allow us to gain information to improve design and conduct of future trials.

DETAILED DESCRIPTION:
This is a ten subject, phase 1 study. The purpose of the study is to demonstrate drug safety in a group with high grade brain tumors and to evaluate cell proliferation with F-18 FLT. FLT is known to clear out of normal brain and detect brain tumor. This population represents a potential clinical population that may benefit from this PET imaging tracer. This information will help improve the design and conduct of future F-18 FLT clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Subject may be male or female and of any race / ethnicity;
* At the time of study drug dosing, the subject has reached his or her 18th birthday;
* Subject has histologic diagnosis of one of the following malignancies - glioblastoma gliosarcoma, anaplastic mixed/anaplastic oligodendroglioma or (anaplastic) astrocytoma with lesion visible on CT or MR and minimum histological grade of III/IV;
* Subject with suspect radiation necrosis that are planned for re-section;
* Subject or subject's legally acceptable representative provides informed consent;
* Subject is capable of complying with study procedures and able to lie still in the PET scanner;
* Subject is capable of communicating with study personnel;
* Subject has adequate liver and kidney function

Exclusion Criteria:

* Subject is pregnant or nursing;
* Subject is anemic (as defined as a hemoglobin level <10);
* Subject has not received chemotherapy or radiation therapy within the two weeks prior to imaging.
* Subject has as reflected by a serum liver enzymes outside the normal laboratory reference range;
* Subject has a history of chronic liver disease, which may compromise liver function;
* Subject has kidney disease as reflected by a serum creatinine outside the normal laboratory reference range;
* Subject has prior history of stroke or other condition of the head or neck that, in the investigator's opinion, might affect circulation to the brain or image interpretation (examples include, but are not limited to, previous stroke with cystic softening and cerebral deformity, or arteriovenous malformation);
* Subject has a history of significant cerebrovascular disease;
* Subject has any other condition or personal circumstance that, in the judgment of the investigator, might interfere with the collection of complete good quality data
* Subject has previously received [F-18]FLT at any time, or any other investigational product within the past two weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-11; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Safety will be demonstrated through analysis of adverse events in subjects enrolled in the trial who received study drug | 24 hr

CONTACTS AND LOCATIONS:
Overall Officials: Charles M Intenzo, MD, Principal Investigator — Thomas Jefferson University Hospital, 132 S 10th St Phila, PA 19107
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States